CLINICAL TRIAL: NCT02594072
Title: Androgen Suppression With Stereotactic Body or External Beam Radiation Therapy (ASSERT): A Phase II Randomized Trial for Intermediate and High Risk Prostate Cancer
Brief Title: Androgen Suppression With Stereotactic Body or External Beam Radiation Therapy (ASSERT)
Acronym: ASSERT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Abraham Alexander, Clinical assistant professor, Radiation Oncologist, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASSERT
Record Dates: First submitted 2015-10-26; First posted 2015-11-02 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SABR with androgen suppression (Experimental): Stereotactic ablative radiotherapy (SABR) with a prescribed dose of 36.25 Gy in 5 fractions over 5 weeks (one treatment day per week). Zoladex ® for androgen suppression, taken for 6 months for patients with intermediate-risk prostate cancer, 18 months for patients with high-risk prostate cancer.
  Interventions: Radiation: stereotactic ablative radiotherapy; Drug: Zoladex ®
- EBRT with androgen suppression (Active Comparator): Conventional external beam radiation therapy (EBRT) with a prescribed dose of 73.68 Gy in 28 fractions (5 treatment days per week over 5.5 weeks). Zoladex ® for androgen suppression, taken for 6 months for patients with intermediate-risk prostate cancer, 18 months for patients with high-risk prostate cancer.
  Interventions: Radiation: external beam radiation therapy; Drug: Zoladex ®

INTERVENTIONS:
Radiation: stereotactic ablative radiotherapy — Linac-based prostate stereotactic radiotherapy, using Volumetric Modulated Arc Therapy planning and delivery, with fiducial marker and cone-beam CT based image guidance.
  Arms: SABR with androgen suppression
Radiation: external beam radiation therapy — Conventional intensity modulated radiotherapy, with fiducial marker or cone-beam CT based image guidance.
  Arms: EBRT with androgen suppression
Drug: Zoladex ® — The preferred agent for the protocol is goserelin acetate (Zoladex ®) 3-month depot, but other LHRH agonists are permitted. The total duration of ADT will be 6 months for men with intermediate risk disease, and 18 months for those with high risk disease. ADT is to be initiated prior to the start of RT.
  Other Names: goserelin acetate

SUMMARY:
Two radiation therapy techniques are commonly used for the treatment of intermediate and high risk prostate cancer: brachytherapy and external beam radiation therapy (EBRT). However, both have limitations. Brachytherapy, in which radioactive seeds are inserted into the prostate, produces excellent outcomes but is invasive and not all patients are eligible or willing to receive this treatment. EBRT, while gentle at the time of delivery, tends to be very prolonged and may have poorer outcomes than brachytherapy. This study will examine the use of stereotactic ablative radiotherapy (SABR), in which patients are given only a few, high dose radiation treatments. Treatments are short, non-invasive, applicable to patients not able to do brachytherapy, and may be more effective than conventional EBRT. This study will compare SABR with EBRT in terms of the rates of acute and late toxicities for each treatment, disease-free survival, and health-related quality of life measures.

DETAILED DESCRIPTION:
The current study is a randomized phase II study comparing high speed, single arc, LINAC-based prostate stereotactic ablative radiotherapy (SABR) with conventional external beam radiation treatment (EBRT), along with androgen suppression (AS), in men with intermediate and high risk prostate cancer, who are either unsuitable for or unwilling to have brachytherapy. The two primary objectives of the study are to assess the feasibility of randomization, and to compare the rates of acute and late toxicities. Should randomization prove feasible, and toxicities comparable, a future phase 3 trial will be pursued.

Primary objectives:

1. To determine the proportion of eligible patients who are willing to be randomized
2. To estimate and compare the proportions of acute and late toxicities, focussing on grade 3 and 4 complications of the treatment interventions as delivered in the British Columbia (BC) Cancer Agency

Secondary objectives:

1. To compare the disease free survival as reflected in biochemical relapse free survival at five years between the two interventions
2. To compare the health related quality of life as reflected in changes on the EPIC questionnaire between the two interventions
3. To quantify the degree of intra-fraction motion with the proposed SABR technique

Research Method

To determine the willingness of eligible patients to be randomized, a screening log documenting the number of eligible subjects approached for participation will be maintained. Subjects who are approached but who decline participation will undergo a short interview by the Clinical Research Associate as to the reason for non-participation. The Clinical Research Associate will read from a script with statements to make sure that subjects who refuse the trial know that they are free to provide or not provide the reasons for declining the trial and that their answers will not affect the care they will receive. They will be asked to list up to five reasons for non-participation in the trial. At the conclusion of the trial, qualitative analyses will be done for the reason of non-participation.

The two radiation treatment protocols, conventional EBRT and SABR, will be compared in a randomized, phase II study.

Patients with biopsy-proven intermediate or high risk prostate cancer will be accrued. T3 or T4 disease, men with International Prostate Symptom Score >20 and prostate volume > 90 cc are not eligible. Men with high risk disease must have a <15% risk of pelvic lymph node involvement to be eligible.

Eligible subjects will be identified by the treating oncologist and enrolled through the clinical trials unit of the participating regional cancer centre. Once the consent form is signed, a Study Entry Form will be sent to the trial administrative centre located at the Vancouver Island Centre of the BC Cancer Agency. A Patient Identification Number will be assigned and the patient will be randomized to a treatment arm. This study proposes that eighty (80) patients be randomized in a 1:1 ratio.

Subjects randomized to Arm 1 (conventional EBRT) will receive 73.68 Gy in 28 fractions (5 treatment days per week over 5.5 weeks).

Subjects randomized to Arm 2 (SABR) will receive a prescribed dose of 36.25 Gy in 5 fractions over 5 weeks (one treatment day per week).

Subjects randomized to the SABR arm will undergo an additional procedure prior to radiation treatment to place gold seed fiducials (placement of gold seed fiducials is optional in the EBRT arm and is at the discretion of the treating centre).

Androgen-Deprivation Therapy (ADT) will be administered to all patients on both treatment arms. ADT will consist of luteinizing hormone-releasing hormone (LHRH) agonist monotherapy, but total androgen blockade is also permitted at the discretion of the treating oncologist. The total duration of ADT will be 6 months for men with intermediate risk disease, and 18 months for those with high risk disease. ADT is to be initiated prior to the start of RT.

PATIENT ASSESSMENTS AND FOLLOWUP

Pre-radiotherapy assessment:

All patients must have a biopsy indicating prostate adenocarcinoma within 365 days of trial registration. A full history and physical examination, with digital rectal examination, must be done within 60 days of registration. CT scan of the abdomen and pelvis and nuclear medicine bone scan must be done within 60 days of registration. Baseline PSA and testosterone must be done not more than 60 days before registration and repeated in the week before radiotherapy to document response to androgen deprivation therapy. Physician assessment must be done within 60 days of randomization. Baseline QOL assessment (EPIC), prostate symptom score (IPSS), and sexual health inventory (SHIM) are to be done prior to the start of radiotherapy.

Assessments during radiotherapy:

All patients will be seen by a radiation oncologist (or clinical associate) weekly during radiotherapy. QOL assessment (EPIC), IPSS/SHIM, and adverse events assessment (CTCAEv4, modified Radiation Therapy Oncology Group (RTOG)/SOMA) will be done during week 5 of radiotherapy for both Arms 1 and 2.

Post-radiotherapy assessment and follow-up:

All patients will be assessed 2 weeks and 8 weeks post-radiotherapy, then every 6 months until 2 years, and then yearly until year 5. At each of these time points patients will undergo physician assessment, PSA/testosterone, QOL assessment (EPIC), IPSS/SHIM, and adverse events assessment (CTCAEv4, modified RTOG/SOMA).

Data Analysis

Actuarial rates of acute (defined as occurring ≤ 6 months after initiation of treatment) and late (defined as occurring > 6 months after initiation of treatment) as well as the prevalence of late toxicities at 1, 2 and 5 years will be determined. Grade 3 and 4 toxicities will be compared between intervention groups using exact test statistics (SAS FREQ procedure, SAS Gary, NC). Stratified analyses will also use the SAS FREQ procedure and Zelen's exact test for equal odds ratios, exact confidence limits for the common odds ratio, and an exact test for the common odds ratio. Quality of life scores and EPIC scales will be compared between interventions using the t-test statistic.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosis of prostate cancer within 365 days prior to registration.
2. Disease must be Canadian Consensus (GUROC) high and intermediate risk with probability of pelvic nodal involvements <15% by the Updated Partin Tables.

   * High risk is defined by any of: ≥T3a, PSA > 20, or Gleason ≥ 8
   * Intermediate risk is defined by: T1/T2 and/or Gleason ≤ 7 and/or PSA ≤20 and not low risk
3. Disease must be T1 or T2 clinically
4. Prostate specific antigen (PSA) and testosterone level (TTT) must be done not more than 60 days before registration. If androgen deprivation therapy is started before registration, PSA and TTT should be done not more than 60 days prior to commencement of androgen deprivation therapy.
5. For high risk patients, negative pelvis CT scan and bone scan for metastases not more than 60 days before registration. If androgen deprivation therapy is started before registration, pelvis CT scan and bone scan should be done not more than 60 days prior to commencement of androgen deprivation therapy. For intermediate risk patients, pelvis CT scan and bone scan are optional.
6. Commencement of androgen deprivation therapy is allowed before registration. However, the lead time must allow for completion of the radiation treatment within 6 months and 18 months of the androgen deprivation therapy treatment duration for intermediate and high risk disease respectively.
7. History/physical examination with digital rectal examination of the prostate within 60 days of registration or commencement of androgen deprivation therapy.
8. Life expectancy of at least 5 years
9. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2
10. No contraindication for 6 months and 18 months of androgen deprivation therapy respectively for intermediate and high risk disease.

Exclusion Criteria:

1. Clinical evidence of extra-prostatic disease extension
2. Clinical evidence of prostate volume > 90 cc prior to randomization
3. Prior history of inflammatory bowel disease
4. Prior history of invasive malignancy (except non-melanomatous skin cancer) or lymphomatous/hematogenous malignancy unless continually disease free for a minimum of 5 years. All patients with in situ carcinoma are eligible for this study (for example, carcinoma in situ of the oral cavity is eligible) except patients with carcinoma of the bladder (including in situ bladder cancer or superficial bladder cancer).
5. Previous pelvic radiation
6. Presence of a hip prosthesis
7. Evidence of pelvic nodal involvement or distant metastases

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-04; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects experiencing treatment-related acute and late toxicities, focussing on grade 3 and 4 complications, as assessed by the NCI CTCAEv4 and modified RTOG/SOMA toxicity scale. | 5 years

SECONDARY OUTCOMES:
Number of subjects with biochemical relapse free survival at five years as measured by PSA levels. | 5 years
To compare the health related quality of life as reflected in changes on the EPIC questionnaire between the two interventions | 5 years
To measure the mean prostate pre-fraction to post-fraction displacement, in millimeters, from CT scans done pre- and post-fraction. | at week 5 of radiotherapy (completion of radiotherapy)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Alexander, MD, Principal Investigator — British Columbia Cancer Agency; Winkle Kwan, MD, Principal Investigator — British Columbia Cancer Agency
Locations (2):
- Canada (2):
  - BC Cancer Agency Fraser Valley Center, Surrey, British Columbia
  - BC Cancer Agency Vancouver Island Center, Victoria, British Columbia